CLINICAL TRIAL: NCT01113125
Title: Topical Treatment With Glucocorticoids to Prevent Hypertrophic Scars and Keloid Due to Central Venous Access in Children
Brief Title: Scars After Central Venous Catheters
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mette Møller Handrup (Other)
Responsible Party: Sponsor-Investigator, Mette Møller Handrup, MD, PhD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-015163-14; 2009-015163-14 (EudraCT Number); 73191198 (Other: Danish Medicines Agency); 20090206 (Other: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Hypertrophic Scars; Keloids
Keywords: hypertrophic scar; keloid; central venous catheter; children; cancer
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid; Neoplasms | interventions — Fusidic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fucicort (Experimental)
  Interventions: Drug: Betamethason-17-valerate and fusidic acid
- Fucidin (Placebo Comparator)
  Interventions: Drug: Fusidic Acid

INTERVENTIONS:
Drug: Betamethason-17-valerate and fusidic acid — 0.4 cm creme is applied and covered with a plaster (treatment under occlusion). Dosage every second or third day Treatment is started one week before removal of the central venous catheter and continued for four weeks
  Arms: Fucicort
Drug: Fusidic Acid — 0.4 cm creme is applied and covered with a plaster (treatment under occlusion). Dosage every second or third day Treatment is started one week before removal of the central venous catheter and continued for four weeks
  Arms: Fucidin

SUMMARY:
Most children with cancer need a central venous catheter. These catheters are typically placed on the anterior thorax, where the risk of hypertrophic scarring and keloid development is greatly enhanced. A significant part of the children who have survived childhood cancer are troubled by their scars.

Topical glucocorticoid treatment is known to induce a reduction of the collagen in the connective tissue.

The investigators hypothesize that treatment with topical glucocorticoids for one week before and three weeks after removal of a central venous catheter, will reduce the formation of hypertrophic scarring and keloid development in children.

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents who have a central venous catheter removed at the Childrens Department of Oncology at Aarhus University Hospital Skejby in the period from March 2010 to July 2011

Exclusion Criteria:

* Known allergy towards plaster or fusidic acid

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-08 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
scars measured by the Vancouver Scar Scale twelve months after central venous catheter removal | Twelve months

SECONDARY OUTCOMES:
Judgement of the scar by Patient and observer scar scale after six months | six months
Judgement of the scar by Patient and observer scar scale after twelve months | twelve months
scars measured by the Vancouver Scar Scale six months after central venous catheter removal | six months

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Hasle, Professor, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Arhus University Hospital Skejby, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Background] Wolfram D, Tzankov A, Pulzl P, Piza-Katzer H. Hypertrophic scars and keloids--a review of their pathophysiology, risk factors, and therapeutic management. Dermatol Surg. 2009 Feb;35(2):171-81. doi: 10.1111/j.1524-4725.2008.34406.x. PMID 19215252
- [Background] Robles DT, Berg D. Abnormal wound healing: keloids. Clin Dermatol. 2007 Jan-Feb;25(1):26-32. doi: 10.1016/j.clindermatol.2006.09.009. PMID 17276198
- [Background] Calaminus G, Weinspach S, Teske C, Gobel U. Quality of survival in children and adolescents after treatment for childhood cancer: the influence of reported late effects on health related quality of life. Klin Padiatr. 2007 May-Jun;219(3):152-7. doi: 10.1055/s-2007-973846. PMID 17525909
- [Background] Sullivan T, Smith J, Kermode J, McIver E, Courtemanche DJ. Rating the burn scar. J Burn Care Rehabil. 1990 May-Jun;11(3):256-60. doi: 10.1097/00004630-199005000-00014. PMID 2373734
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Hopwood P, Fletcher I, Lee A, Al Ghazal S. A body image scale for use with cancer patients. Eur J Cancer. 2001 Jan;37(2):189-97. doi: 10.1016/s0959-8049(00)00353-1. PMID 11166145